CLINICAL TRIAL: NCT01106326
Title: A Pilot Study to Improve Preventive Asthma Care for Urban Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 28198
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Teens participating in this study will have:
  1. directly observed administration of their daily preventive asthma medication at school, by the school nurse, for the first 6-8 weeks of the study
  2. three counseling sessions with a study nurse trained in principles of motivational interviewing (MI), that are designed to enhance the teen's motivation to change health behaviors, with a focus on adherence to evidence-based preventive care guidelines (e.g.; preventive medications).
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Teens participating in this study will have:
  1. directly observed administration of their daily preventive asthma medication at school, by the school nurse, for the first 6-8 weeks of the study
  2. three counseling sessions with a study nurse trained in principles of motivational interviewing (MI), that are designed to enhance the teen's motivation to change health behaviors, with a focus on adherence to evidence-based preventive care guidelines (e.g.; preventive medications).

SUMMARY:
The goal of this pilot study is to implement directly observed therapy with preventive asthma medications through a partnership with the school nurse (with input and direction from the primary care provider) to assure that the teen receives guideline based preventive medications, and provide a motivational interviewing intervention to help the teen transition to independence with their medical treatment plan. We hypothesize that this community-based pilot intervention will; 1) be feasible and acceptable among this population and among school personnel, and 2) yield reduced asthma morbidity (symptom-free days, absenteeism, and emergency room / urgent care use for asthma care). We anticipate that enhancing preventive healthcare for urban teens with asthma through partnerships with schools will yield improved health, prevention of suffering, decreased absenteeism from school, and reduced healthcare costs. This new method of preventive care delivery could be sustained within the school nursing system, and could be implemented in schools nationwide. Further, it could be applied to other chronic illnesses affecting disadvantaged populations.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma
* Persistent asthma (criteria based on NHLBI guidelines).
* Age >12 and <15 years.
* Attending school in the Rochester City School District.
* Signed physician permission to enroll the child.
* Current prescription of a daily preventive asthma medication
* Parent or caregiver and the adolescent must consent to the intervention.

Exclusion Criteria:

* Inability to speak and understand English.
* No access to a working phone for follow-up surveys
* The family planning to leave the school district within fewer than 6 months.
* The teen having other significant medical conditions
* The teen having a diagnosed developmental condition per parent report.
* Adolescents in foster care or other situations in which consent cannot be obtained from a guardian.
* Adolescents that were previously enrolled in our School-Based Asthma Study

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Blaakman SW, Cohen A, Fagnano M, Halterman JS. Asthma medication adherence among urban teens: a qualitative analysis of barriers, facilitators and experiences with school-based care. J Asthma. 2014 Jun;51(5):522-9. doi: 10.3109/02770903.2014.885041. Epub 2014 Feb 7. PMID 24494626
- [Result] Halterman JS, Riekert K, Bayer A, Fagnano M, Tremblay P, Blaakman S, Borrelli B. A pilot study to enhance preventive asthma care among urban adolescents with asthma. J Asthma. 2011 Jun;48(5):523-30. doi: 10.3109/02770903.2011.576741. PMID 21599562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptom-free Days Over Two Weeks
Description: We will measure number of symptom-free days at 2-months (at the end of the directly observed therapy phase) and 4-months (after their transition to independence with preventive medications). We anticipate that teens will experience more symptom-free days compared to baseline assessment.
Time Frame: 2 and 4 month follow-up assessments
Population: Analysis conducted per protocol.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Baseline | Two Months Post Baseline | Four Months Post Baseline
Number analyzed (Participants) | 30 | 28 | 28
Days | 10.79 (3.74) | 8.71 (4.66) | 12.89 (1.62)

2. Secondary Outcome: Additional Asthma Morbidity Measures
Description: We also will compare additional baseline asthma morbidity measures, quality of life, health care utilization, cotinine, and exhaled nitric oxide with outcomes at the follow-up assessments.
Time Frame: 2 month, 4 month, final follow-up assessments
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No